CLINICAL TRIAL: NCT01291394
Title: Easypod Connect: A National, Multicentre, Observational Registry to Study Adherence and Long Term Outcomes of Therapy in Paediatric Subjects Using Easypod™ Electromechanical Device for Growth Hormone Treatment
Brief Title: To Assess the Level of Adherence of Subjects Receiving SAIZEN® Via Easypod™ in France
Acronym: ECOS FRA
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200104-515
Record Dates: First submitted 2011-01-31; First posted 2011-02-08 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Growth Disorders
Keywords: Growth disorders; Saizen; Easypod; Growth hormone; Pediatric subject
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Easypod™ — Saizen (Somatotropin) as per Summary of Product Characteristics administered by Easypod™
  Other Names: Somatotropin

SUMMARY:
This is a National, Multicentre, Observational Registry to study adherence and long term outcomes of therapy in paediatric subjects using Easypod™ electromechanical device for growth hormone treatment from hospitals in France and to assess the level of adherence of subjects receiving SAIZEN® via Easypod™.

DETAILED DESCRIPTION:
Subjects will be enrolled in this observational, multi-center study to assess adherence and treatment outcomes. Parents will provide their written agreement to upload their child's data in the study electronic CRF.

Easypod™ is an electromechanical device that delivers growth hormone and also records injections' date and time. Adherence data will be primarily derived from injections recorded in the Easypod™ device combined with physician data entry of outcome measures (i.e. height & weight). This will allow the establishment of adherence profiles and evaluate the link with subsequent clinical outcomes.

Since this is an observational study, there will be no study-specific clinical interventions and subjects will be treated according to the clinical and laboratory findings as routinely evaluated by the physician. Auxological and laboratory data will be reported prospectively throughout the duration of the study. At baseline, available data can be recorded retrospectively from the subjects' medical file and Easypod™ device Data will be collected retrospectively and prospectively. This will allow the establishment of adherence profiles and subsequent clinical outcomes. Collected data will be also analyzed in a multinational pooled analysis of comparable national studies.

Primary Objective:

• To assess the level of adherence of subjects receiving Saizen® via Easypod™

Secondary Objectives:

* To describe the impact of adherence on clinical outcomes for subject receiving Saizen® via Easypod™
* To identify adherence subject profiling
* To asses the Impact of adherence on insulin-like growth factor-1 (IGF1) ranges/levels

ELIGIBILITY:
Inclusion Criteria:

* Administered Saizen® via the Easypod™ electromechanical device according to pediatric registered indications (Growth Hormone Deficiency, Small for Gestational Age, Turner-Syndrome or prepubertal children with Chronic Renal Failure).
* Naïve subjects or already treated with Saizen and Easypod for maximum 1 year
* Male and Female between 2 - 18 years of age, or over 18 without fusion of growth plates
* Parent's or guardian's (or subject if over 18 without fusion of growth plates) written agreement, given before entering data into the study, with the understanding that the subject or parent/guardian may withdraw agreement at any time without prejudice to future medical care.

Exclusion Criteria:

* Subjects taking Saizen® in whom growth plates have fused (i.e. taking growth hormone for it's metabolic effects)
* Contra-indications to Saizen® as defined in the French Summary of Product Characteristics (SmPC)
* Use of an investigational drug or participation in an interventional clinical study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who are taking SAIZEN® for a pediatric registered indications using the Easypod™ electromechanical device.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2011-01-31 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mean percent of recorded adherence | At least 6 months and up to 5 years

SECONDARY OUTCOMES:
Correlation of adherence and growth outcome (change in height velocity (HV), change in HV-Standard Deviation Score (HV-SDS), change in height-Standard Deviation Score) after each year of Saizen® treatment with Easypod™ | At least 6 months and up to 5 years
Subject adherence profile | At least 6 months and up to 5 years
  Subject adherence profile based on age, gender, indication, self-injection or not, time on treatment, administration regimen (6 or 7 days/ week), combination of pituitary hormone deficiencies, previous and/or concomitant treatments, socio-economic data
Correlation of adherence with IGF-1 levels/ranges | At least 6 months and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MGS Division, Merck Serono s.a.s, France, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Contact Merck KGaA, Communication Center, France

REFERENCES:
- [Result] Koledova, E. et al. (2017) Analysis of results from the global, 5-year Easypod™ Connect Observational Study (ECOS) study in children with growth disorders. 10th International Meeting for Pediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Result] Wit, JM. et al. (2017) Effect of adherence on the 2-year growth response to growth hormone treatment in prepubertal children with idiopathic isolated growth hormone deficiency participating in the EasypodTM Connect Observational Study (ECOS). 10th International Meeting of Paediatric Endocrinology; 2017 Sep 14-17; Washington, DC.